CLINICAL TRIAL: NCT03034187
Title: Radiation Induced Toxicity in Prostate Cancer
Brief Title: Radiation-induced Toxicity in Prostate Cancer/ Standard-Follow-Up Program Prostate
Acronym: SFP-PROSTATE
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: H1998-12/SFP-Prostate
Record Dates: First submitted 2016-09-27; First posted 2017-01-27 (Estimated); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Prostate Cancer
Keywords: Acute toxicity; Late toxicity; Quality of Life since 2011(set-up SFP-prostate)
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal is to gain insight in the development and course of the toxicity after a curative treatment of prostate cancer

DETAILED DESCRIPTION:
All with curative intent treated prostate cancer patients will be enrolled in the SFP (Standard Follow-up Programme). It also includes the post -operative adjuvant treatments and the patients with positive lymph nodes.

Patients will complete weekly questionnaires to score the patient -rated toxicity. Biweekly patients are seen by the treating radiation oncologist and / or AIOS in which the physician -rated toxicity is scored. In the follow-up will always patient -rated toxicity and physician -rated toxicity can be determined.

Use of an SFP should yield a profit for the practitioner , such as the automatic generation of letters. This should apply to all SFPs .

Quality of life and toxicity in patients will be completed on the touch-screen computers at FU visits.

ELIGIBILITY:
Inclusion Criteria:

* All curative treated patients with prostatecancer( with positive lymph nodes)
* All patients who will be treated with RT( including post-operative, adjuvant treatments)
* Are willing to fill in toxicity and QOL-questionnarys (QLQ-PR25 en de QLQ-C30)

Exclusion Criteria:

Patients who are not willing to fill in toxicity and QOL-questionnarys Patients who will not get RT Non-curative or palliative treated patients (with bone mestasis) Non-prostate cancer-patients

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All with curative intent treated prostate cancer patients who will be treated with RT will be enrolled in the SFP.
  It also includes the post-surgical adjuvant treatment and patients with positive lymph nodes to research the development and toxicity after RT
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 1999-04; Primary Completion 2025-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
1. Change in Acute toxicity | Toxicity:First visit/Wekely during RT, Acute Toxicity: 2-wekely and at the end of RT/ 2 months after RT/1, 2, 3, 4, 5 years after RT
  Common Terminology Criteria for Adverse Events, version 4.0
  * CTCAE 4.0 Constipation
  * CTCAE 4.0 Diarrhea
  * CTCAE 4.0 Fecal Incontinence
  * CTCAE 4.0 Flatulance
  * CTCAE 4.0 Proctitis
  * CTCAE 4.0 Rectal Hemorrhage
  * CTCAE 4.0 Rectal Mucositis
  * CTCAE 4.0 Rectal Ulcer
  * CTCAE 4.0 Bladder spasm
  * CTCAE 4.0 Cystitis Noninfective
  * CTCAE 4.0 Hematuria
  * CTCAE 4.0 Urinary Frequency
  * CTCAE 4.0 Urinary Incontinence
  * CTCAE 4.0 Urinary retention
  * CTCAE 4.0 Urinary tract Obstruction
  * CTCAE 4.0 Urinary tract pain
  * CTCAE 4.0 Urinary Urgency
  * CTCAE 4.0 Erectile dysfunction

SECONDARY OUTCOMES:
2. Change in patient -rated Quality-of-Life | First visit/End of RT/ 2 months after RT/1, 2, 3, 4, 5 years after RT
  Questionnarys QLQ-PR25, QLQ-C30, International Index of Erectile Function

OTHER OUTCOMES:
3. Change in physiological parameters | First visit/2 months after RT/1, 2, 3, 4, 5 years after RT
  PSA and Testosteron
4. Change in Acute/ Late toxicity(physician rated) | First Visit/ 2 wekely/ End of RT/ 2 months after RT/1, 2, 3, 4, 5 years after RT
  Common Terminology Criteria for Adverse Events, version 4.0
  * CTCAE 4.0 Constipation
  * CTCAE 4.0 Diarrhea
  * CTCAE 4.0 Fecal Incontinence
  * CTCAE 4.0 Flatulance
  * CTCAE 4.0 Proctitis
  * CTCAE 4.0 Rectal Hemorrhage
  * CTCAE 4.0 Rectal Mucositis
  * CTCAE 4.0 Rectal Ulcer
  * CTCAE 4.0 Bladder spasm
  * CTCAE 4.0 Cystitis Noninfective
  * CTCAE 4.0 Hematuria
  * CTCAE 4.0 Urinary Frequency
  * CTCAE 4.0 Urinary Incontinence
  * CTCAE 4.0 Urinary retention
  * CTCAE 4.0 Urinary tract Obstruction
  * CTCAE 4.0 Urinary tract pain
  * CTCAE 4.0 Urinary Urgency
  * CTCAE 4.0 Erectile dysfunction

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Sharing data between physicians at the Department of Radiotherapy